CLINICAL TRIAL: NCT02196701
Title: Concomitant Longitudinal Evaluation of Adalimumab With Methotrexate in the Real World: the CLEAR Study
Acronym: CLEAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: W14-406
Record Dates: First submitted 2014-07-18; First posted 2014-07-22 (Estimated); Results first posted 2018-03-19 (Actual); Last update posted 2018-03-19 (Actual); Status verified 2018-01

CONDITIONS: Psoriasis
Keywords: methotrexate; adalimumab; biologic; psoriasis; Tumor necrosis factor (TNF)-α inhibitor
MeSH Terms: conditions — Psoriasis | interventions — Adalimumab; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adalimumab Plus Methotrexate (Experimental): Participants received 40 mg adalimumab every other week and methotrexate, between 7.5 and 25 mg/week at the discretion of the Investigator, for 24 weeks.
  Interventions: Drug: Adalimumab; Drug: Methotrexate

INTERVENTIONS:
Drug: Adalimumab — Administered by subcutaneous injection every other week.
  Other Names: Humira
Drug: Methotrexate — Methotrexate was provided as 2.5 mg tablets for oral administration.

SUMMARY:
The purpose of this study is to determine the safety and efficacy of the use of the combination therapy adalimumab (ADA) every other week (EOW) with methotrexate (MTX) in suboptimal responders to ADA monotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have been on ADA monotherapy (40 mg eow or greater) for at least 16 weeks but who in the opinion of the Investigator have shown a sub-optimal response to treatment and have a Physician's Global Assessment (PGA) of ≥ 3 and a Psoriasis Area Severity Index (PASI) of ≥ 5; or Subjects who after an initial positive response to ADA monotherapy (40 mg eow or greater) have failed to maintain an optimal level of response, based on the opinion of the Investigator, and have a PGA of ≥ 3 and a PASI of ≥ 5;
2. Subjects who are receiving 40 mg ADA once weekly must be on ADA 40 mg eow for 8 weeks prior to screening;
3. Subjects with at least a 6 month history of chronic plaque psoriasis;
4. Subjects greater than or equal to 18 years of age;
5. If female, subject is either not of childbearing potential, defined as postmenopausal for at least 1 year or surgically sterile or is of childbearing potential and is practicing birth control;
6. The results of the serum pregnancy test performed during the Screening Period and urine pregnancy test performed at the Baseline Visit must be negative;
7. Subject is judged to be in good general health as determined by the Principal Investigator;
8. Subjects must be evaluated for latent tuberculosis (TB) infection;
9. Subjects must be able and willing to provide written informed consent and comply with the requirements of the study protocol;
10. Subjects must be willing and able to self-administer subcutaneous (SC) injections or have a qualified person available to administer SC injections.

Exclusion Criteria:

1. Subject has any contraindications to MTX or ADA;
2. Subject has a previous failed response or poor tolerance to ADA;
3. Subject has a poorly controlled medical condition which, in the opinion of the Investigator, would put the subject at risk by participation in the study;
4. Subject has a history of clinically significant hematologic, renal or liver disease;
5. Subject has a history of neurologic symptoms suggestive of central nervous system (CNS) demyelinating disease and/or diagnosis of central demyelinating disease;
6. Subject has evidence of dysplasia or history of malignancy (including lymphoma and leukemia) other than a successfully treated non-metastatic cutaneous squamous cell or basal cell carcinoma or localized carcinoma in situ of the cervix;
7. Subject has a history of listeriosis, histoplasmosis, untreated TB, persistent chronic infections, or recent active infections requiring hospitalization or treatment with intravenous (iv) anti-infectives within 30 days or oral anti-infectives within 14 days prior to the Baseline visit;
8. Subject is known to have immune deficiency, history of human immunodeficiency virus (HIV) or is immunocompromised;
9. Subject currently uses or plans to use anti-retroviral therapy at any time during the study;
10. Female subject who is pregnant or breast-feeding or considering becoming pregnant during the study or for 150 days after the last dose of study medication;
11. Subject has a history of clinically significant drug or alcohol usage in the last year or cannot maintain an alcohol intake of 30 g a day or less throughout the study (one standard drink is defined as 180 mL/6 oz (approx. 10 g) of wine, 360 mL/12 oz (approx. 15 g) of regular beer, or 45 mL/1.5 oz (approx. 10 g) of spirits;
12. Screening clinical laboratory analyses show any of the following abnormal laboratory results:

    * Aspartate transaminase (AST) or alanine transaminase (ALT) > 2x the upper limit of normal (ULN);
    * Serum total bilirubin > 1.5 mg/dL (> 26 micromol/L), except for subjects with Gilbert's Syndrome;
    * Creatinine > 1.5 mg/dL (133 micromol/L) in subjects ≤ 65 years old and > upper limit of normal range in subjects > 65;
    * Positive Hepatitis B or C serology indicative of previous or current infection.
13. Subject is considered by the Investigator, for any reason, to be an unsuitable candidate for the study;
14. The following treatments are prohibited for all subjects during the study:

    * Phototherapy (ultraviolet A with psoralen [PUVA] within 4 weeks of the Baseline Visit and/or ultraviolet B (UVB) within 2 weeks of the Baseline Visit);
    * Other biologic therapies (including any other anti-tumor necrosis factor [TNF]) within 4 weeks of the Baseline Visit;
    * Any investigational agents of chemical or biologic nature within a minimum of 30 days or 5 half-lives (whichever is longer) of the drug prior to the Baseline visit ;
    * Any other systemic drug therapies for psoriasis within 4 weeks of the Baseline Visit;
    * Oral or injectable corticosteroids, new prescription topical therapies, or changes in the concentration of current prescription topical therapies (including corticosteroids) that are being used, within 2 weeks of the Baseline Visit. Subjects may continue using previously prescribed topical therapies (including corticosteroids) during the study.
15. Prior exposure to biologics that have a potential or known association with progressive multifocal leukoencephalopathy (PML), i.e., natalizumab (Tysabri®) or rituximab (Rituxan®);
16. Subjects with any active viral infection that based on the investigator's clinical assessment makes the subject an unsuitable candidate for the study;

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2014-08-05 (Actual); Primary Completion 2017-03-17 (Actual); Study Completion 2017-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc-André Raymond, PhD, Study Director — AbbVie

REFERENCES:
- See also: Related Info — http://rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This single-arm, open-label longitudinal study was conducted at 12 sites in Canada from 5 August 2014 to 17 March 2017. The study entailed a screening period up to 35 days, a 24-week treatment period, and a 70-day safety follow-up period. Participants continued to receive adalimumab (ADA) and had oral methotrexate (MTX) added to their treatment.
Pre-assignment Details: This study enrolled participants who in the opinion of the Investigator were not responding optimally to adalimumab monotherapy at least 16 weeks after initiating treatment (primary sub-optimal responders) or who after an initial positive response to ADA monotherapy failed to maintain an optimal level of response (secondary sub-optimal responders).
Groups:
- Adalimumab + Methotrexate: Participants received 40 mg adalimumab every other week and methotrexate, between 7.5 and 25 mg/week at the discretion of the Investigator, for 24 weeks.
Period: Overall Study
Arm/Group | Adalimumab + Methotrexate
Started | 46
Completed | 43
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Lost to Follow-up | 1
Not completed — Non-adherence to Protocol | 1

BASELINE CHARACTERISTICS:
Groups:
- Primary Sub-optimal Responders - ADA + MTX: Participants who did not respond optimally to ADA monotherapy at least 16 weeks after initiating treatment (primary sub-optimal responders) received 40 mg adalimumab every other week and methotrexate, between 7.5 and 25 mg/week at the discretion of the Investigator, for 24 weeks.
- Secondary Sub-optimal Responders - ADA + MTX: Participants who after an initial positive response to ADA monotherapy failed to maintain an optimal level of response (secondary sub-optimal responders) received 40 mg adalimumab every other week and methotrexate, between 7.5 and 25 mg/week at the discretion of the Investigator, for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Primary Sub-optimal Responders - ADA + MTX | Secondary Sub-optimal Responders - ADA + MTX | Total
Number analyzed (Participants) | 6 | 40 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (13.84) | 47.3 (11.91) | 46.5 (12.20)
Age, Customized [Count of Participants; unit: Participants]
  < 40 years | 2 | 13 | 15
  40 - 64 years | 4 | 22 | 26
  ≥ 65 years | 0 | 5 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 9 | 11
  Male | 4 | 31 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 39 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 31 | 35
  Black | 0 | 1 | 1
  Asian | 2 | 8 | 10
Duration of Psoriasis [Mean (Standard Deviation); unit: years] | 20.623 (10.4819) | 21.760 (9.7403) | 21.612 (9.7253)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a Satisfactory Response at Week 16 Based on Investigator Assessment
Description: Study investigators were asked to complete the following questionnaire at week 16:
  Overall, at this point in time, how satisfied are you with the psoriasis control provided by the subject's current treatment regimen? The response choices provided were:
  * Completely dissatisfied
  * Moderately dissatisfied
  * Slightly satisfied
  * Highly satisfied
  * Completely satisfied
  Satisfaction with therapy was defined by the combination of highly or completely satisfied responses.
Time Frame: Week 16
Population: Participants who received at least one dose of ADA and one dose of MTX. Participants with missing values at week 16 were categorized as non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Sub-optimal Responders - ADA + MTX | Secondary Sub-optimal Responders - ADA + MTX | Adalimumab + Methotrexate
Number analyzed (Participants) | 6 | 40 | 46
percentage of participants | 33.3 [0.0 to 71.1] | 52.5 [37.0 to 68.0] | 50.0 [35.6 to 64.4]

2. Primary Outcome: Percentage of Participants Achieving a Satisfactory Response at Week 16 Based on Patient Self-assessment
Description: Participants were asked to complete the following questionnaire at week 16:
  Overall, at this point in time, how satisfied are you with your current treatment for psoriasis? The response choices provided were:
  * Completely dissatisfied
  * Moderately dissatisfied
  * Slightly satisfied
  * Highly satisfied
  * Completely satisfied
  Satisfaction with therapy was defined by the combination of highly or completely satisfied responses.
Time Frame: Week 16
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Sub-optimal Responders - ADA + MTX | Secondary Sub-optimal Responders - ADA + MTX | Adalimumab + Methotrexate
Number analyzed (Participants) | 6 | 40 | 46
percentage of participants | 16.7 [0.0 to 46.5] | 52.5 [37.0 to 68.0] | 47.8 [33.4 to 62.3]

3. Secondary Outcome: Percentage of Participants Achieving a Satisfactory Response Based on Investigator Assessment Over Time
Description: Study investigators were asked to complete the following questionnaire at each scheduled visit:
  Overall, at this point in time, how satisfied are you with the psoriasis control provided by the subject's current treatment regimen? The response choices provided were:
  * Completely dissatisfied
  * Moderately dissatisfied
  * Slightly satisfied
  * Highly satisfied
  * Completely satisfied
  Satisfaction with therapy was defined by the combination of highly or completely satisfied responses.
Time Frame: Baseline, week 8 and week 24
Population: Participants who received at least one dose of ADA and one dose of MTX. Participants with missing values were categorized as non-responders.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Sub-optimal Responders - ADA + MTX | Secondary Sub-optimal Responders - ADA + MTX | Adalimumab + Methotrexate
Number analyzed (Participants) | 6 | 40 | 46
percentage of participants
  Baseline | 0 [0.0 to 0.0] | 0 [0.0 to 0.0] | 0 [0.0 to 0.0]
  Week 8 | 50.0 [10.0 to 90.0] | 42.5 [27.2 to 57.8] | 43.5 [29.2 to 57.8]
  Week 24 | 33.3 [0.0 to 71.1] | 60.0 [44.8 to 75.2] | 56.5 [42.2 to 70.8]

4. Secondary Outcome: Percentage of Participants Achieving a Satisfactory Response Based on Patient Self-assessment Over Time
Description: Participants were asked to complete the following questionnaire at each scheduled visit:
  Overall, at this point in time, how satisfied are you with your current treatment for psoriasis? The response choices provided were:
  * Completely dissatisfied
  * Moderately dissatisfied
  * Slightly satisfied
  * Highly satisfied
  * Completely satisfied
  Satisfaction with therapy was defined by the combination of highly or completely satisfied responses.
Time Frame: Baseline, week 8 and week 24
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Sub-optimal Responders - ADA + MTX | Secondary Sub-optimal Responders - ADA + MTX | Adalimumab + Methotrexate
Number analyzed (Participants) | 6 | 40 | 46
percentage of participants
  Baseline | 0 [0.0 to 0.0] | 17.5 [5.7 to 29.3] | 15.2 [4.8 to 25.6]
  Week 8 | 16.7 [0.0 to 46.5] | 52.5 [37.0 to 68.0] | 47.8 [33.4 to 62.3]
  Week 24 | 16.7 [0.0 to 46.5] | 60.0 [44.8 to 75.2] | 54.3 [40.0 to 68.7]

5. Secondary Outcome: Number of Participants Achieving Each Satisfactory Category Based on Investigator Assessment Over Time
Description: Study investigators were asked to complete the following questionnaire at each scheduled visit:
  Overall, at this point in time, how satisfied are you with the psoriasis control provided by the subject's current treatment regimen? The response choices provided were:
  * Completely dissatisfied
  * Moderately dissatisfied
  * Slightly satisfied
  * Highly satisfied
  * Completely satisfied
Time Frame: Baseline, weeks 8, 16, and 24
Population: Participants who received at least one dose of ADA and one dose of MTX with available data at each time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab + Methotrexate
Number analyzed (Participants) | 46
Participants
  Baseline: Completely satisfied | 0
  Baseline: Highly satisfied | 0
  Baseline: Slightly satisfied | 8
  Baseline: Moderately dissatisfied | 31
  Baseline: Completely dissatisfied | 7
  Baseline: Missing | 0
  Week 8: Completely satisfied | 6
  Week 8: Highly satisfied | 14
  Week 8: Slightly satisfied | 15
  Week 8: Moderately dissatisfied | 9
  Week 8: Completely dissatisfied | 1
  Week 8: Missing | 1
  Week 16: Completely satisfied | 8
  Week 16: Highly satisfied | 15
  Week 16: Slightly satisfied | 10
  Week 16: Moderately dissatisfied | 8
  Week 16: Completely dissatisfied | 3
  Week 16: Missing | 2
  Week 24: Completely satisfied | 11
  Week 24: Highly satisfied | 15
  Week 24: Slightly satisfied | 7
  Week 24: Moderately dissatisfied | 6
  Week 24: Completely dissatisfied | 4
  Week 24: Missing | 3

6. Secondary Outcome: Number of Participants Achieving Each Satisfactory Category Based on Patient Self-assessment Over Time
Description: Participants were asked to complete the following questionnaire at each scheduled visit:
  Overall, at this point in time, how satisfied are you with your current treatment for psoriasis? The response choices provided were:
  * Completely dissatisfied
  * Moderately dissatisfied
  * Slightly satisfied
  * Highly satisfied
  * Completely satisfied
Time Frame: Baseline, weeks 8, 16, and 24
Population: Participants who received at least one dose of ADA and one dose of MTX and with available data at each time point..
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab + Methotrexate
Number analyzed (Participants) | 46
Participants
  Baseline: Completely satisfied | 5
  Baseline: Highly satisfied | 2
  Baseline: Slightly satisfied | 15
  Baseline: Moderately dissatisfied | 17
  Baseline: Completely dissatisfied | 7
  Baseline: Missing | 0
  Week 8: Completely satisfied | 10
  Week 8: Highly satisfied | 12
  Week 8: Slightly satisfied | 14
  Week 8: Moderately dissatisfied | 7
  Week 8: Completely dissatisfied | 2
  Week 8: Missing | 1
  Week 16: Completely satisfied | 7
  Week 16: Highly satisfied | 15
  Week 16: Slightly satisfied | 13
  Week 16: Moderately dissatisfied | 6
  Week 16: Completely dissatisfied | 3
  Week 16: Missing | 2
  Week 24: Completely satisfied | 10
  Week 24: Highly satisfied | 15
  Week 24: Slightly satisfied | 7
  Week 24: Moderately dissatisfied | 6
  Week 24: Completely dissatisfied | 5
  Week 24: Missing | 3

7. Secondary Outcome: Percentage of Participants Who Achieved a Psoriasis Area and Severity Index (PASI) 50 Response Over Time
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The PASI score ranges from 0 (no psoriasis) to 72 (very severe psoriasis). A PASI 50 response is defined as at least a 50% reduction (improvement) from baseline in PASI score.
Time Frame: Baseline and Weeks 8, 16, and 24
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Sub-optimal Responders - ADA + MTX | Secondary Sub-optimal Responders - ADA + MTX | Adalimumab + Methotrexate
Number analyzed (Participants) | 6 | 40 | 46
percentage of participants
  Week 8 | 50.0 [10.0 to 90.0] | 42.5 [27.2 to 57.8] | 43.5 [29.2 to 57.8]
  Week 16 | 50.0 [10.0 to 90.0] | 62.5 [47.5 to 77.5] | 60.9 [46.8 to 75.0]
  Week 24 | 66.7 [28.9 to 100.0] | 65.0 [50.2 to 79.8] | 65.2 [51.5 to 79.0]

8. Secondary Outcome: Percentage of Participants Who Achieved a PASI 75 Response Over Time
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The PASI score ranges from 0 (no psoriasis) to 72 (very severe psoriasis). A PASI 75 response is defined as at least a 75% reduction (improvement) from baseline in PASI score.
Time Frame: Baseline and Weeks 8, 16, and 24
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Sub-optimal Responders - ADA + MTX | Secondary Sub-optimal Responders - ADA + MTX | Adalimumab + Methotrexate
Number analyzed (Participants) | 6 | 40 | 46
percentage of participants
  Week 8 | 33.3 [0.0 to 71.1] | 27.5 [13.7 to 41.3] | 28.3 [15.2 to 41.3]
  Week 16 | 16.7 [0.0 to 46.5] | 42.5 [27.2 to 57.8] | 39.1 [25.0 to 53.2]
  Week 24 | 16.7 [0.0 to 46.5] | 42.5 [27.2 to 57.8] | 39.1 [25.0 to 53.2]

9. Secondary Outcome: Percentage of Participants Who Achieved a PASI 90 Response Over Time
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The PASI score ranges from 0 (no psoriasis) to 72 (very severe psoriasis). A PASI 90 response is defined as at least a 90% reduction (improvement) from baseline in PASI score.
Time Frame: Baseline and Weeks 8, 16, and 24
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Sub-optimal Responders - ADA + MTX | Secondary Sub-optimal Responders - ADA + MTX | Adalimumab + Methotrexate
Number analyzed (Participants) | 6 | 40 | 46
percentage of participants
  Week 8 | 16.7 [0.0 to 46.5] | 12.5 [2.3 to 22.7] | 13.0 [3.3 to 22.8]
  Week 16 | 16.7 [0.0 to 46.5] | 15.0 [3.9 to 26.1] | 15.2 [4.8 to 25.6]
  Week 24 | 16.7 [0.0 to 46.5] | 30.0 [15.8 to 44.2] | 28.3 [15.2 to 41.3]

10. Secondary Outcome: Percentage of Participants Who Achieved a PASI 100 Response Over Time
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The PASI score ranges from 0 (no psoriasis) to 72 (very severe psoriasis). A PASI 100 response is defined as a 100% reduction (improvement) from baseline in PASI score.
Time Frame: Baseline and Weeks 8, 16, and 24
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Sub-optimal Responders - ADA + MTX | Secondary Sub-optimal Responders - ADA + MTX | Adalimumab + Methotrexate
Number analyzed (Participants) | 6 | 40 | 46
percentage of participants
  Week 8 | 16.7 [0.0 to 46.5] | 12.5 [2.3 to 22.7] | 13.0 [3.3 to 22.8]
  Week 16 | 16.7 [0.0 to 46.5] | 10.0 [0.7 to 19.3] | 10.9 [1.9 to 19.9]
  Week 24 | 16.7 [0.0 to 46.5] | 27.5 [13.7 to 41.3] | 26.1 [13.4 to 38.8]

11. Secondary Outcome: Change From Baseline in PASI Score Over Time
Description: PASI is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (plaque thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The PASI score ranges from 0 (no psoriasis) to 72 (very severe psoriasis).
Time Frame: Baseline and weeks 8, 16, and 24
Population: Participants who received at least one dose of ADA and one dose of MTX. A mixed-effect model repeat measurement was used.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Primary Sub-optimal Responders - ADA + MTX | Secondary Sub-optimal Responders - ADA + MTX | Adalimumab + Methotrexate
Number analyzed (Participants) | 6 | 40 | 46
units on a scale
  Week 8: number analyzed (Participants) | 6 | 39 | 45
  Week 8 | -4.6 (2.07) | -4.6 (0.65) | -4.6 (0.61)
  Week 16: number analyzed (Participants) | 6 | 38 | 44
  Week 16 | -4.5 (1.31) | -6.2 (0.59) | -5.9 (0.53)
  Week 24: number analyzed (Participants) | 6 | 37 | 43
  Week 24 | -3.1 (3.17) | -6.3 (0.68) | -5.9 (0.74)

12. Secondary Outcome: Percent Change From Baseline in PASI Score
Description: as for outcome 11
Time Frame: Baseline and weeks 8, 16, and 24
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Primary Sub-optimal Responders - ADA + MTX | Secondary Sub-optimal Responders - ADA + MTX | Adalimumab + Methotrexate
Number analyzed (Participants) | 6 | 40 | 46
percent change
  Week 8: number analyzed (Participants) | 6 | 39 | 45
  Week 8 | -51.6 (16.23) | -43.7 (6.11) | -44.8 (5.64)
  Week 16: number analyzed (Participants) | 6 | 38 | 44
  Week 16 | -45.6 (15.15) | -59.2 (5.06) | -57.3 (4.74)
  Week 24: number analyzed (Participants) | 6 | 37 | 43
  Week 24 | -17.4 (45.65) | -63.7 (5.78) | -58.1 (8.01)

13. Secondary Outcome: Percentage of Participants Achieving a Physician's Global Assessment of Disease Activity (PGA) of Cleared or Minimal Over Time
Description: The PGA is a 6-point scale used to measure the severity of disease at the time of the evaluation. The degree of overall lesion severity was evaluated using the following categories:
  * 0 (Cleared): No evidence of scaling, erythema, or plaque elevation;
  * 1 (Minimal): Occasional fine scale over <5% of lesions, faint erythema, minimal plaque elevation;
  * 2 (Mild): Fine scale dominates, light red coloration, mild plaque elevation;
  * 3 (Moderate): Course scale dominates, moderate red coloration, moderate plaque elevation;
  * 4 (Marked): Thick non-tenacious scale dominates, bright red coloration, marked plaque elevation;
  * 5 (Severe): Very thick tenacious scale predominates, dusky to deep red coloration, severe plaque elevation.
  The percentage of participants achieving a score of clear (0) or minimal (1) is reported.
Time Frame: Weeks 8, 16, and 24
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Sub-optimal Responders - ADA + MTX | Secondary Sub-optimal Responders - ADA + MTX | Adalimumab + Methotrexate
Number analyzed (Participants) | 6 | 40 | 46
percentage of participants
  Week 8 | 16.7 [0.0 to 46.5] | 27.5 [13.7 to 41.3] | 26.1 [13.4 to 38.8]
  Week 16 | 16.7 [0.0 to 46.5] | 35.0 [20.2 to 49.8] | 32.6 [19.1 to 46.2]
  Week 24 | 16.7 [0.0 to 46.5] | 47.5 [32.0 to 63.0] | 43.5 [29.2 to 57.8]

14. Secondary Outcome: Change From Baseline in Body Surface Area (BSA) Affected by Psoriasis
Description: The total body surface area affected by psoriasis (expressed as a percentage) was measured by the investigator using the palm method, where the participant's hand represents 1% of body surface area.
  A decrease in BSA affected by psoriasis indicates improvement.
Time Frame: Baseline and weeks 8, 16, and 24
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: percentage of body surface area
Arm/Group | Primary Sub-optimal Responders - ADA + MTX | Secondary Sub-optimal Responders - ADA + MTX | Adalimumab + Methotrexate
Number analyzed (Participants) | 6 | 40 | 46
percentage of body surface area
  Week 8: number analyzed (Participants) | 5 | 39 | 44
  Week 8 | -3.5 (2.95) | -4.5 (1.06) | -4.4 (0.98)
  Week 16: number analyzed (Participants) | 6 | 38 | 44
  Week 16 | -4.5 (2.40) | -6.4 (1.08) | -6.2 (0.99)
  Week 24: number analyzed (Participants) | 6 | 37 | 43
  Week 24 | -4.1 (1.57) | -6.3 (0.89) | -6.0 (0.79)

15. Secondary Outcome: Percent Change From Baseline in Body Surface Area (BSA) Affected by Psoriasis
Description: as for outcome 14
Time Frame: Baseline and weeks 8, 16, and 24
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Primary Sub-optimal Responders - ADA + MTX | Secondary Sub-optimal Responders - ADA + MTX | Adalimumab + Methotrexate
Number analyzed (Participants) | 6 | 40 | 46
percent change
  Week 8: number analyzed (Participants) | 5 | 39 | 44
  Week 8 | -33.9 (23.10) | -34.1 (7.48) | -33.4 (7.17)
  Week 16: number analyzed (Participants) | 6 | 38 | 44
  Week 16 | -34.1 (22.25) | -54.2 (5.89) | -51.4 (5.89)
  Week 24: number analyzed (Participants) | 6 | 37 | 43
  Week 24 | -32.7 (22.25) | -61.7 (6.33) | -57.8 (6.21)

16. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) Score Over Time
Description: The DLQI questionnaire asks participants to evaluate the degree that psoriasis has affected their quality of life in the last week, and includes the following parameters: symptoms and feelings, daily activities, leisure activities, work or school activities, personal relationships and treatment related feelings. Participants answer 10 questions on a scale from 0 (not at all) to 3 (very much); the range of the total score is 0 to 30. A score of 21 to 30 means an extremely large effect on the participant's life whereas 0-1 means that the disease has no effect at all. A negative change from Baseline indicates improvement.
Time Frame: Baseline, weeks 8, 16, and 24
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Primary Sub-optimal Responders - ADA + MTX | Secondary Sub-optimal Responders - ADA + MTX | Adalimumab + Methotrexate
Number analyzed (Participants) | 6 | 40 | 46
units on a scale
  Week 8: number analyzed (Participants) | 6 | 39 | 45
  Week 8 | -5.0 (1.40) | -4.8 (0.71) | -4.8 (0.64)
  Week 16: number analyzed (Participants) | 6 | 38 | 44
  Week 16 | -3.8 (2.54) | -5.9 (0.78) | -5.6 (0.76)
  Week 24: number analyzed (Participants) | 6 | 37 | 43
  Week 24 | -1.7 (4.29) | -6.3 (0.69) | -5.4 (0.88)

17. Secondary Outcome: Percent Change From Baseline in Dermatology Life Quality Index (DLQI) Score Over Time
Description: as for outcome 16
Time Frame: Baseline, weeks 8, 16, and 24
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Primary Sub-optimal Responders - ADA + MTX | Secondary Sub-optimal Responders - ADA + MTX | Adalimumab + Methotrexate
Number analyzed (Participants) | 6 | 40 | 46
percent change
  Week 8: number analyzed (Participants) | 6 | 39 | 45
  Week 8 | -43.0 (21.50) | -38.6 (7.01) | -39.2 (6.48)
  Week 16: number analyzed (Participants) | 6 | 38 | 44
  Week 16 | -22.9 (40.40) | -38.9 (12.79) | -36.7 (11.85)
  Week 24: number analyzed (Participants) | 6 | 37 | 43
  Week 24 | 14.4 (71.98) | -55.0 (6.90) | -44.5 (11.11)

18. Secondary Outcome: Percentage of Participants Who Achieved a DLQI Score of 0 or 1 Over Time
Description: The DLQI questionnaire asks participants to evaluate the degree that psoriasis has affected their quality of life in the last week, and includes the following parameters: symptoms and feelings, daily activities, leisure activities, work or school activities, personal relationships and treatment related feelings. Participants answer 10 questions on a scale from 0 (not at all) to 3 (very much); the range of the total score is 0 to 30. A score of 21 to 30 means an extremely large effect on the participant's life whereas 0-1 means that the disease has no effect at all.
Time Frame: Baseline and Weeks 8, 16, and 24
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Primary Sub-optimal Responders - ADA + MTX | Secondary Sub-optimal Responders - ADA + MTX | Adalimumab + Methotrexate
Number analyzed (Participants) | 6 | 40 | 46
percentage of participants
  Week 8 | 16.7 [0.0 to 46.5] | 20.0 [7.6 to 32.4] | 19.6 [8.1 to 31.0]
  Week 16 | 16.7 [0.0 to 46.5] | 40.0 [24.8 to 55.2] | 37.0 [23.0 to 50.9]
  Week 24 | 16.7 [0.0 to 46.5] | 40.0 [24.8 to 55.2] | 37.0 [23.0 to 50.9]

19. Secondary Outcome: Change From Baseline in High-sensitivity C-reactive Protein (Hs-CRP) at Week 24
Time Frame: Baseline and week 24
Population: as for outcome 11
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Primary Sub-optimal Responders - ADA + MTX | Secondary Sub-optimal Responders - ADA + MTX | Adalimumab + Methotrexate
Number analyzed (Participants) | 6 | 39 | 45
mg/L | -2.6 (0.47) | 0.1 (1.52) | -0.3 (1.32)

ADVERSE EVENTS:
Time Frame: From the date of either the first dose of study adalimumab or the first dose of methotrexate up to 70 days after the last adalimumab injection during the study. The median duration of exposure to adalimumab was 168 days (range: 14 - 171 days).
Arm/Group | Adalimumab + Methotrexate
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 1/46
Other Adverse Events (participants affected / at risk) | 27/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab + Methotrexate (N=46)
Cardiac arrest (Cardiac disorders) | 1
Generalised tonic-clonic seizure (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adalimumab + Methotrexate (N=46)
Vision blurred (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Chest pain (General disorders) | 1
Cyst (General disorders) | 1
Fatigue (General disorders) | 2
Vessel puncture site bruise (General disorders) | 1
Beta haemolytic streptococcal infection (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 3
Folliculitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 7
Pharyngitis streptococcal (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 2
Streptococcal bacteraemia (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 2
Tooth infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 2
Lower limb fracture (Injury, poisoning and procedural complications) | 1
Seroma (Injury, poisoning and procedural complications) | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 1
Liver function test increased (Investigations) | 1
Gout (Metabolism and nutrition disorders) | 2
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Polymyalgia rheumatica (Metabolism and nutrition disorders) | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1
Neuralgia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 2
Mood altered (Psychiatric disorders) | 1
Sleep disorder (Psychiatric disorders) | 1
Crystalluria (Renal and urinary disorders) | 1
Vulvovaginal dryness (Reproductive system and breast disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 2
Hypotension (Vascular disorders) | 1
Peripheral venous disease (Vascular disorders) | 1
Dizziness (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2016-04-22): https://cdn.clinicaltrials.gov/large-docs/01/NCT02196701/Prot_000.pdf
  • Statistical Analysis Plan (2017-03-29): https://cdn.clinicaltrials.gov/large-docs/01/NCT02196701/SAP_001.pdf